CLINICAL TRIAL: NCT00656305
Title: A Pivotal Study to Evaluate the Effectiveness and Safety of ExAblate Treatment of Metastatic and Multiple Myeloma Bone Tumors for the Palliation of Pain in Patients Who Are Not Candidates for Radiation Therapy
Brief Title: ExAblate (MRgFUS) Treatment of Metastatic Bone Tumors for the Palliation of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BM004
Record Dates: First submitted 2008-04-02; First posted 2008-04-11 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Bone Metastases; Multiple Myeloma
Keywords: Bone Cancer; Pain Palliation; Metastasis; Multiple Myeloma; Breast Cancer; Lung Cancer; Prostate Cancer; cancer related Pain; Tumors
MeSH Terms: conditions — Multiple Myeloma; Bone Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Cancer Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- ExAblate Treatment Arm (Experimental)
  Interventions: Device: ExAblate MRfFUS
- ExAblate Sham Arm (Sham Comparator)
  Interventions: Device: ExAblate MRfFUS; Device: Sham

INTERVENTIONS:
Device: ExAblate MRfFUS — MR guided focused ultrasound.
  Other Names: MRgFUS; FUS; Focused Ultrasound; MR guided Focused Ultrasound
Device: Sham — sham comparator
  Arms: ExAblate Sham Arm

SUMMARY:
A Pivotal Study to Evaluate the Effectiveness and Safety of ExAblate Treatment of Metastatic Bone and Multiple Myeloma Tumors for the Palliation of Pain in Patients Who are not Candidates for Radiation Therapy

ELIGIBILITY:
Inclusion criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are suffering from symptoms of bone metastases or multiple myeloma bone lesions and are radiation failure patients:

   Radiation failure candidates are those who have received radiation without adequate relief from metastatic bone pain as determined by the patient and treating physician, those for whom their treating physician would not prescribe radiation or additional radiation treatments, and those patients who refuse additional radiation therapy,
4. Patients who refuse other accepted available treatments such as surgery or narcotics for pain alleviation.
5. Patient with NRS (0-10 scale) pain score ≥ 4 irrespective of medication
6. Targeted tumor(s) are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5)
7. Targeted tumor (treated) size up to 55 cm2 in surface area
8. Patient whose targeted (treated) lesion is on bone and the interface between the bone and lesion is deeper than 10-mm from the skin.
9. Targeted (treated) tumor clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible
10. Able to communicate sensations during the ExAblate treatment
11. Patients on ongoing chemotherapy regimen for at least 1 month at the time of eligibility:

    - with same chemotherapy regimen (as documented from patient medical dossier),

    And

    - Worst pain NRS still >= 4

    And

    - do NOT plan to initiate a new chemotherapy for pain palliation should be eligible for the study.
12. No radiation therapy to targeted (most painful) lesion in the past two weeks
13. Bisphosphonate intake should remain stable throughout the study duration.
14. Patients will have from 1 to 5 painful lesions and only the most painful lesion will be treated.
15. Patients with persistent distinguishable pain associated with 1 site to be treated (if patient has pain from additional sites, the pain from the additional sites must be evaluated as being less intense by at least 2 points on the NRS compared to the site to be treated).

Exclusion Criteria:

1. Patients who either

   * Need surgical stabilization of the affected bony structure (>7 fracture risk score, see Section 7.3) OR
   * Targeted tumor is at an impending fracture site (>7 on fracture risk score, see Section 7.3).

   OR

   - Patients with surgical stabilization of tumor site with metallic hardware
2. More than 5 painful lesions, or more than 1 requiring immediate localized treatment
3. Targeted (treated) tumor is in the skull
4. Patients on dialysis
5. Patients with life expectancy < 3-Months
6. patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
7. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication
   * Patients with documented myocardial infarction within six months of protocol entry
   * Congestive heart failure requiring medication (other than diuretic)
   * Patients on anti-arrhythmic drugs
8. Severe hypertension (diastolic BP > 100 on medication)
9. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations (weight >250 pounds), etc.
10. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
11. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
12. KPS Score < 60 (See "Definitions" below)
13. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
14. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
15. Target (treated) tumor is less then 1cm from nerve bundles, bowels or bladder.
16. Are participating or have participated in another clinical trial in the last 30 days
17. Patients initiating a new chemotherapy regime, or radiation (for the targeted most painful lesion) within the last 2 weeks
18. Patients unable to communicate with the investigator and staff.
19. Patients with persistent undistinguishable pain (pain source unidentifiable)
20. Targeted (treated) tumor surface area >= 55 cm2
21. Patient whose bone-lesion interface is < 10-mm from the skin
22. Targeted (treated) tumor NOT visible by non-contrast MRI,
23. Targeted (most painful) tumor Not accessible to ExAblate
24. The targeted tumor is less than 2 points more painful compared to other painful lesions on the site specific NRS.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (8):
  - University of California San Diego, La Jolla, California
  - Stanford University Medical Center, Stanford, California
  - University MRI & Diagnostic Imaging Centers, Boca Raton, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
- Toronto General Hospital, Toronto, Ontario, Canada
- Israel (2):
  - Rambam medical Center -The Pain palliation unit, Haifa
  - Sheba Medical Center, Tel Litwinsky
- University of Rome "La Sapienza", Rome, Italy
- Russia (2):
  - Rostov State Research Institute of Oncology, Rostov-on-Don
  - N. N. Petrov Institute of Oncology, Saint Petersburg

REFERENCES:
- [Derived] Bitton RR, Rosenberg J, LeBlang S, Napoli A, Meyer J, Butts Pauly K, Hurwitz M, Ghanouni P. MRI-Guided Focused Ultrasound of Osseous Metastases: Treatment Parameters Associated With Successful Pain Reduction. Invest Radiol. 2021 Mar 1;56(3):141-146. doi: 10.1097/RLI.0000000000000721. PMID 32858582
- [Derived] Hurwitz MD, Ghanouni P, Kanaev SV, Iozeffi D, Gianfelice D, Fennessy FM, Kuten A, Meyer JE, LeBlang SD, Roberts A, Choi J, Larner JM, Napoli A, Turkevich VG, Inbar Y, Tempany CM, Pfeffer RM. Magnetic resonance-guided focused ultrasound for patients with painful bone metastases: phase III trial results. J Natl Cancer Inst. 2014 Apr 23;106(5):dju082. doi: 10.1093/jnci/dju082. PMID 24760791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 147 subjects enrolled (signed consent), 23 subjects failed additional study requirements and 9 subjects exited after randomization but prior to treatment
Groups:
- ExAblate Treatment Arm: ExAblate 2000: MR guided focused ultrasound
- ExAblate Sham Control Arm: ExAblate 2000: MR guided focused ultrasound sham
Period: Overall Study
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm
Started | 87 | 28
Completed | 65 | 21
Not Completed | 22 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm | Total
Number analyzed (Participants) | 87 | 28 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.3) | 56.8 (10.5) | 57.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 22 | 71
  Male | 38 | 6 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 81 | 26 | 107
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 1 | 7
  United States | 30 | 11 | 41
  Italy | 0 | 1 | 1
  Israel | 17 | 5 | 22
  Russia | 34 | 10 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: Using the Numerical Rating Score (NRS) for pain (0 being no pain and 10 being worst imaginable pain), each subject was rated as a Responder or Non-responder. A responder is defined as a subject with a reduction in NRS worst score from baseline of two (2) or more points, and no increase in pain medication use.
Time Frame: 3 months post treatment
Population: 115 subjects were underwent treatment. Of these, 4 subjects terminated treatment prior to full completion. These 4 subjects are excluded from the efficacy analysis. An additional 4 subjects were found to have been enrolled in the study more than once. In a pre-PMA meeting with FDA, it was agreed upon to exclude these 4 subjects from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm
Number analyzed (Participants) | 81 | 26
Participants | 54 | 6

2. Secondary Outcome: Number of Participants With a Change in Medication Use
Description: Medication Use change reported from baseline until of study. Medication use is quantified by "morphine equivalent usage" (measured separately from Responder/Non-responder definition for the primary endpoint)
Time Frame: 3 months post treatment
Population: Only 26 of the 81 subjects in ExAblate treatment arm and 6 of 26 in the sham arm were taking non-opioid medication at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm
Number analyzed (Participants) | 26 | 6
Participants | 15 | 2

3. Secondary Outcome: Quality of Life (QOL) as Measured by Change in Bodily Pain Inventory (BPI) From Baseline
Description: The BPI-QOL questionnaire is designed to show the severity and interference of pain in the lives of patients. This is a 7-item questionnaire that asks respondents the extent to which pain interferes with their general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life using a 0-10 numerical rating scale in which 0 represents 'does not interfere' and 10 indicates 'completely interferes'. Responses to the 7 items are averaged to form the pain interference scale score. Lower scores are better, showing less interference in daily activities while higher scores show more interference and hence worse outcomes.
Time Frame: 3 months post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm
Number analyzed (Participants) | 81 | 26
score on a scale | 2.5 (2.8) | .3 (2.3)

ADVERSE EVENTS:
Arm/Group | ExAblate Treatment Arm | ExAblate Sham Control Arm
All-Cause Mortality (participants affected / at risk) | 8/87 | 0/28
Serious Adverse Events (participants affected / at risk) | 8/87 | 0/28
Other Adverse Events (participants affected / at risk) | 49/87 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ExAblate Treatment Arm (N=87) | ExAblate Sham Control Arm (N=28)
Death (Immune system disorders) | 8 | 0 — 8 subjects died due to cancer progression, unrelated to study procedures.
Hospitalization (Surgical and medical procedures) | 1 | 0 — Transient congnitive decline observed pre treatment resulting in gamma knife resection of brain metastasis.
Hospitalization (Surgical and medical procedures) | 1 | 0 — Surgery for fracture at ExAblate-treatment site
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment Arm (N=87) | ExAblate Sham Control Arm (N=28)
Deep Vein Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Skin burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy/leg pain (Nervous system disorders) | 2 (2) | 0 (0)
Pain/discomfort (Injury, poisoning and procedural complications) | 46 (48) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No